CLINICAL TRIAL: NCT03598673
Title: The Efficacy and Tolerability of Highly Selective Beta-1 Agent in Hypertensive Black Patients Residing in Sub Saharan Africa: A Pilot Study
Brief Title: To Determine the Effect of Nebivolol on Office Blood Pressure of Blacks Residing in Nigeria
Acronym: Nevibolol
Status: Completed | Type: Observational
Sponsor: University of Abuja (Other)
Collaborators: Micronova Pharmaceuticals Ind Ltd (Unknown)
Responsible Party: Principal Investigator, Dr. Dike Ojji, Principal Investigator, University of Abuja
Other Study IDs: UAbuja
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertensives to receiving Nevibolol: Patients to receive Nevibolol
  Interventions: Drug: The Efficacy and Tolerability of Nebivolol in Nigerians

INTERVENTIONS:
Drug: The Efficacy and Tolerability of Nebivolol in Nigerians — To determine the effect of Nevibolol on office blood pressure of Blacks residing in Nigeria
  Other Names: Effect of Nebivolol in Nigeria

SUMMARY:
Although Nebivolol, a highly selective beta-1 agent has been shown to be effective in reducing blood pressure in Blacks, this was in African Americans with no study in Blacks residing in sub Saharan Africa. We therefore decided to study the effectiveness and safety of Nebivolol in Black patients with stage 1 hypertension (systolic BP of 140-149 and/or diastolic BP of 90-99 mmHg) presenting to five primary care centres in Nigeria.

DETAILED DESCRIPTION:
Although Nebivolol, a highly selective beta-1 agent has been shown to be effective in reducing blood pressure in Blacks, this was in African Americans with no study in Blacks residing in sub Saharan Africa. It might be argued that findings in African-Americans can be extrapolated to Black Africans since they have the same ancestral origin, the differences in selection in previous generations, ethnic admixture and differences in lifestyle suggest that such an extrapolation may be inappropriate. We are therefore studying the effectiveness and safety of Nebivolol in Black patients with stage 1 hypertension (systolic BP of 140-149 and/or diastolic BP of 90-99 mmHg) presenting to primary care centres in Nigeria.

We hypothesise based on previous findings of the effect of Nebivolol on blood control of African Americans, we hypothesise that 5mg and 10mg of Nebivolol will be effective and well tolerated by black hypertensive patients residing in Nigeria.

The primary objective is to study the effect of 5mg and 10mg of Nebivolol on blood pressure control in Black African hypertensive patients residing in Nigeria. The secondary objectives are: to evaluate the rates of BP control (<140 mmHg systolic and <90 mmHg diastolic) achieved with 5mg and 10mg of Nebivolol respectively; to evaluate the incidence and the nature of adverse events with these two doses of Nebivolol; to evaluate the effects of these two doses of Nebivolol on fasting blood sugar and fasting lipid profile, and to evaluate the effect of these two doses on erectile dysfunction The primary outcome measure is change in office BP value from baseline to 2 months. This will be calculated as the difference between the mean office BP at randomization and that at the end of follow up. And the secondary endpoints are: to determine the proportion of patients who achieve BP <140 mmHg systolic and <90 mmHg diastolic in two months; to determine the proportion of patients who have adverse events with both doses of Nebivolol respectively; to study the change in plasma fasting blood sugar and fasting lipid profile over two months, and to see proportion of male patients who complain of erectile dysfunction on follow up and end of the study.

It is is a prospective, observational program among hypertensive patients with 3 months follow up.

ELIGIBILITY:
Inclusion Criteria: The patients should be aged 30-59 years with a sitting SBP ≥140 mm Hg and <160 mmHg and/or DBP ≥ 90 and <100 mmHg on no antihypertensive agent

Exclusion Criteria:

1.Those with clinically defined congestive heart failure 2. Those with clinical features of renal failure 3. Those with history of coronary heart disease including chronic stable angina, myocardial infarction or acute coronary syndrome 4. Patients with a history of a stroke or transient ischaemic attack 5. Patients with known or suspected secondary hypertension 6. Those with any other concomitant illness, physical or mental impairment that could interfere with the effective conduct of the study 7. Those who are pregnant or those of child-bearing age who are not taking reliable contraception.

-

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients should be aged 30-59 years with a sitting SBP ≥140 mm Hg and <160 mmHg and/or DBP ≥ 90 and <100 mmHg on no antihypertensive agent.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2019-04-27 (Actual)

PRIMARY OUTCOMES:
Change in office blood pressure | 2 months
  The primary outcome measure is change in office BP value from baseline to 2 months

SECONDARY OUTCOMES:
The proportion of patients who achieved blood control | 2 months
  The proportion of patients who achieved BP <140 mmHg systolic and <90 mmHg diastolic in two months.
Proportion of patients with adverse events | 1 month and 2 months
  The proportion of patients who have adverse events with both doses of Nebivolol respectively
Change in metabolic profile | 2 months
  Change in plasma fasting blood sugar and fasting lipid profile over two months.
Proportion of male patients with erectile dysfunction | 1 month and 2 months
  The proportion of male patients who complain of erectile dysfunction on follow up and end of the study

CONTACTS AND LOCATIONS:
Locations (2):
- Nigeria (2):
  - Africa International College, Abuja, Federal Capital Territory
  - University of Abuja Teaching Hospital, Abuja, Federal Capital Territory

REFERENCES:
- [Derived] Ojji D, Ale BM, Shedul L, Umuerri E, Ejim E, Alikor C, Agunyenwa C, Njideofor U, Eze H, Ansa V. The Effect of Nebivolol on Office Blood Pressure of Blacks Residing in Sub-Saharan Africa (A Pilot Study). Front Cardiovasc Med. 2021 Jan 11;7:613917. doi: 10.3389/fcvm.2020.613917. eCollection 2020. PMID 33505995